CLINICAL TRIAL: NCT04149379
Title: Hyperbaric Oxygen Therapy After Cerebral Infarction - PILOT
Brief Title: Hyperbaric Oxygen Therapy After Stroke - PILOT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of the economic consequences of the COVID-19 pandemic 2020
Sponsor: Norwegian Underwater Intervention (NUI) (Industry)
Collaborators: Western Norway University of Applied Sciences (Other); Helse-Bergen HF (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 305476
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Stroke
Keywords: Stroke; Hyperbaric oxygen
MeSH Terms: conditions — Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Single subject SSED
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): One group of 6 patients undergoing 20 sessions of hyperbaric therapy at table 14/90.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — 20 sessions of hyperbaric therapy in a pressure chamber at 2,4 absolute atmospheres, 90 minutes per day of breathing 100% medical oxygen through an own mask. Table 14/90.

SUMMARY:
The goal of this pilot study is to establish more information about hyperbaric oxygen therapy for this group of patients, and give us more information of how to initiate the best possible main study. Can we find any indications that support the use of this therapy for patients suffering from chronic disability after cerebral infarction? Can we improve physical and cognitive function.

DETAILED DESCRIPTION:
This is a pilot project including 6 patients for one session of 20 treatments of hyperbaric oxygen therapy. The objective is to establish knowledge of HBO for this group of patients in a Norwegian context, so that we can prepare for the main study afterwards, including about 60-70 patients. We need to know how to optimize the administrative and technical systems for the larger study. We want to collect feedback from the patients undergoing the pilot study. We want more information about the treatment table, if 20 treatments are enough, if 2,4 bar pressure is adequate. The treatment table is based on existing research, and is considered safe.

The patients are to be treated at table 14/90, at 2,4 Absolute atmospheres, and daly 90 minutes of oxygen inhalation (medical oxygen).

ELIGIBILITY:
Inlcution criteria:

* No age restriction
* Suffered from ischemic stroke (cerebral infarction) 6-12 months before inclusion.
* Stable phase after standard rehabilitation
* Measurable physical function failure and / or reduced ADL function.
* Sufficient physical function / mobility to be able to move into / out of the pressure chamber with the help of only one person (Tender).

Patients to participate in the study must be physically, mentally and cognitively fit for pressure chamber treatment. They must be able to stand for their own help, move with support, and be able to follow instructions. This is ensured by discretionary assessment after observation and interview with the patient.

Exclusion criteria:

* Claustrophobia
* Psychosis, severe anxiety
* Inability to equalize pressure in the middle ear
* Severe COPD and asthma, pathological lung sounds
* Hypertension (Blood pressure > 140/90 mmHg)
* Pregnancy
* Hernia
* Earlier fractures, or suspected fractures in the face
* Ongoing chemotherapy
* Previous treatment with Bleomycin
* Aphasia that prevents necessary communication
* Cognitive failure that prevents necessary co-operation in the pressure chamber.
* Previous or current pneumothorax, other lung injury
* Increased risk of pneumothorax

  * Known or suspected injury to the chest
  * Marfan syndrome
  * Homocystinuria
  * Family history of pneumothorax
  * Chronic lung disease (COPD, Emphysema, Asthma eller cystic fibrosis)
  * Tuberculosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Improved physical and cognitive function in activities of daily living. | 0+6+12 months after end of treatment period
  The project's physiotherapist and ergo therapist from Western Norway University of Applied Sciences (HVL) are responsible for examining physical function and the participant's ability to acquire and use knowledge, as well as function in everyday living activities (ADL). Three measurements are made before starting treatment (establishing a baseline), where the third measurement is done on the same day as treatment starts to eliminate changes in test results as a result of learning the tests. Measurements are also made immediately after the end of treatment, as well as follow-up measurements after 6 and 12 months. Descriptions below.
Short Physical Performance Battery (SPPB) | 0+6+12 months after end of treatment period
  This test is very widely used to provide a quick and validated test of strength, balance and coordination. The test has a roof effect, so it is not suitable for capturing very small and subtle self-perceived disturbances in function. The test is very sensitive to change in the target group.
Grip strength | 0+6+12 months after end of treatment period
  There is a recognized and validated connection between general function and health and grip strength, as well as between grip strength and life span. Grip strength changes as other function changes.
Fatigue Severity Scale (FSC) | 0+6+12 months after end of treatment period
  A major problem after stroke and in many brain disorders is fatigue. Fatigue leads to reduced foxing and thus loss of function. The test is believed to be able to detect changes that are relevant to everyday life function and social participation.
Canadian Occupational Performance Measure (COPM) | 0+6+12 months after end of treatment period
  COPM is designed to help people identify and prioritize activity problems, as well as evaluate activity performance and satisfaction with activity execution. In an interview, the person is asked to describe activities they consider important but find it difficult to perform. Among the aforementioned challenges, the person is asked to prioritize a maximum of five activities he / she wants to be able to perform better after the end of treatment. Then, the person is asked to score the current performance and satisfaction with the current performance of priority activities. The score scale is from 1-10 where 10 indicates very good workmanship or high satisfaction. After the interview, partial scores for execution (COPM-U) and satisfaction (COPM-T) are calculated. A change score of 3 points is considered a clinically important change. COPM has shown good measurement properties, among other things for participants with stroke and the elderly.
Action Research Arm Test (ARAT) | 0+6+12 months after end of treatment period
  ARAT is a tool designed to assess motor function in the arm after stroke. The tasks in the test reflect daily activities and the patient's ability to perform them. The test contains 19 sub-tasks in which different grips (five-finger grips, cylinder grips, tweezers grips), as well as gross motor skills are specifically assessed. In each of the 19 tasks, a score is given from 0-3, where high scores indicate good arm function. The total score (0-57) is the sum of the sub-scores. The test has shown promising measurement properties. For participants in the chronic and subacute phase after stroke, a change of 5.7 points (10%) is considered clinically important. Norwegian guidelines will be used in the study.
Nine Hole Peg Test (NHPT) | 0+6+12 months after end of treatment period
  NHPT is a simple test of fine motor skills that is recommended, among other things, for participants with stroke. Scoring is based on the time the patient spends in placing and removing nine small pieces in nine holes. Total time (maximum 50 seconds) and total number of pins are indicated. The test has shown satisfactory reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Tobba T Südmann, PhD, Principal Investigator — Western Norway University of Applied Sciences
Locations (1):
- NUI, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heyboer M 3rd, Sharma D, Santiago W, McCulloch N. Hyperbaric Oxygen Therapy: Side Effects Defined and Quantified. Adv Wound Care (New Rochelle). 2017 Jun 1;6(6):210-224. doi: 10.1089/wound.2016.0718. PMID 28616361
- [Background] Plafki C, Peters P, Almeling M, Welslau W, Busch R. Complications and side effects of hyperbaric oxygen therapy. Aviat Space Environ Med. 2000 Feb;71(2):119-24. PMID 10685584
- [Background] Mu J, Ostrowski RP, Soejima Y, Rolland WB, Krafft PR, Tang J, Zhang JH. Delayed hyperbaric oxygen therapy induces cell proliferation through stabilization of cAMP responsive element binding protein in the rat model of MCAo-induced ischemic brain injury. Neurobiol Dis. 2013 Mar;51:133-43. doi: 10.1016/j.nbd.2012.11.003. Epub 2012 Nov 10. PMID 23146993
- [Result] Mathieu D, Marroni A, Kot J. Tenth European Consensus Conference on Hyperbaric Medicine: recommendations for accepted and non-accepted clinical indications and practice of hyperbaric oxygen treatment. Diving Hyperb Med. 2017 Mar;47(1):24-32. doi: 10.28920/dhm47.1.24-32. PMID 28357821
- [Result] Al-Waili NS, Butler GJ, Beale J, Abdullah MS, Hamilton RW, Lee BY, Lucus P, Allen MW, Petrillo RL, Carrey Z, Finkelstein M. Hyperbaric oxygen in the treatment of patients with cerebral stroke, brain trauma, and neurologic disease. Adv Ther. 2005 Nov-Dec;22(6):659-78. doi: 10.1007/BF02849960. PMID 16510383
- [Result] Efrati S, Ben-Jacob E. Reflections on the neurotherapeutic effects of hyperbaric oxygen. Expert Rev Neurother. 2014 Mar;14(3):233-6. doi: 10.1586/14737175.2014.884928. Epub 2014 Jan 29. PMID 24471697
- [Result] Rosario ER, Kaplan SE, Khonsari S, Vazquez G, Solanki N, Lane M, Brownell H, Rosenberg SS. The Effect of Hyperbaric Oxygen Therapy on Functional Impairments Caused by Ischemic Stroke. Neurol Res Int. 2018 Oct 9;2018:3172679. doi: 10.1155/2018/3172679. eCollection 2018. PMID 30402285
- [Result] Wang W, Osenbroch P, Skinnes R, Esbensen Y, Bjoras M, Eide L. Mitochondrial DNA integrity is essential for mitochondrial maturation during differentiation of neural stem cells. Stem Cells. 2010 Dec;28(12):2195-204. doi: 10.1002/stem.542. PMID 20954243
- [Result] Efrati S, Fishlev G, Bechor Y, Volkov O, Bergan J, Kliakhandler K, Kamiager I, Gal N, Friedman M, Ben-Jacob E, Golan H. Hyperbaric oxygen induces late neuroplasticity in post stroke patients--randomized, prospective trial. PLoS One. 2013;8(1):e53716. doi: 10.1371/journal.pone.0053716. Epub 2013 Jan 15. PMID 23335971
- [Result] Godman CA, Chheda KP, Hightower LE, Perdrizet G, Shin DG, Giardina C. Hyperbaric oxygen induces a cytoprotective and angiogenic response in human microvascular endothelial cells. Cell Stress Chaperones. 2010 Jul;15(4):431-42. doi: 10.1007/s12192-009-0159-0. Epub 2009 Dec 1. PMID 19949909
- [Result] Vila JF, Balcarce PE, Abiusi GR, Dominguez RO, Pisarello JB. Improvement in motor and cognitive impairment after hyperbaric oxygen therapy in a selected group of patients with cerebrovascular disease: a prospective single-blind controlled trial. Undersea Hyperb Med. 2005 Sep-Oct;32(5):341-9. PMID 16457083
- See also: The effects of combined hyperbaric oxygen therapy on patients with post-stroke depression — https://www.jstage.jst.go.jp/article/jpts/27/5/27_jpts-2014-730/_article/-char/ja/